CLINICAL TRIAL: NCT03175042
Title: Non-invasive Spot Hemoglobin Measurement in the Outpatient Obstetric Clinic
Status: Completed | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 17-0095
Record Dates: First submitted 2017-05-31; First posted 2017-06-05 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2018-04

CONDITIONS: Anemia in Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Pregnant patients with anemia: Pregnant patients meeting Center for Disease Control (CDC) guidelines for anemia during pregnancy will be screened for participation in the study. In the outpatient setting at our institution it is standard of care that these women have complete blood counts (CBCs) drawn every 4-6 weeks. At the time of the routine blood draw, we will place the non invasive monitor on their finger to record the hemoglobin value. We will be comparing the hemoglobin values obtained from the CBC to that obtained from the non-invasive monitor.
  Interventions: Device: Masimo spot hemoglobin non-invasive monitor

INTERVENTIONS:
Device: Masimo spot hemoglobin non-invasive monitor — This non-invasive monitor measures hemoglobin using LED light technology. We will be using it to determine if it is as accurate as routine CBC in anemic obstetric patients.

SUMMARY:
Pregnant patients in the UT Medical Branch outpatient obstetric clinic are screened for anemia via blood draw at first prenatal visit. Those who meet Center for Disease Control (CDC) criteria for anemia during pregnancy (hemoglobin less than 11g/dL in first and third trimesters and hemoglobin less than 10.5g/dL during the second trimester), will be approached for participation in this study. It is the protocol of the UT Medical Branch outpatient obstetric clinic to repeat a blood draw every 4 weeks in patients with anemia. At the time of their blood draw, patients who participate in our study will have the Masimo Spot Non-invasive Hemoglobin monitor placed on our finger. The primary aim of the study is to see how accurate the non-invasive monitor is compared with blood draw. With the potential benefit being earlier diagnosis of anemia and easier method to ensure improvement in the hemoglobin.

DETAILED DESCRIPTION:
Pregnant women who are patients in the UT Medical Branch outpatient obstetric clinic will be screened for anemia using blood draw for CBC during the first prenatal visit. Those who are found to have anemia will be prospectively enrolled in this proof-of-concept study. Anemia will be defined according to the CDC guidelines (first and third trimesters hemoglobin level less than 11g/dL, and less than 10.5g/dL in the second trimester). Patients meeting these criteria will be approached for inclusion. If patients consent to participate, they will have their hemoglobin checked via the non-invasive monitor at the same time as their clinically indicated CBC testing. At the UT Medical Branch outpatient obstetric clinic, this is usually every 3-4 weeks and determined by the health care provider. The hemoglobin measured by the non-invasive monitor will be compared with the hemoglobin obtained via the complete blood count. Other data collected from the patient's medical record will include general characteristics such as demographics, medical history and hemoglobin levels obtained from blood draw.

ELIGIBILITY:
Inclusion Criteria:

pregnant women aged 18-50 with anemia (hemoglobin less than 11g/dL during first and third trimester and less than 10.5g/dL during second trimester)

Exclusion Criteria:

patients with normal hemoglobin levels patients with hemoglobinopathy (sickle cell disease) patients who are incarcerated patients unwilling or unable to give consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant patients, aged 18-50, in the UTMB Outpatient Obstetric Clinic with anemia (defined as hemoglobin less than 11g/dL during first and third trimester and less than 10.5g/dL during second trimester)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Hemoglobin values | During pregnancy (maximum 40 weeks)
  Comparing hemoglobin values between CBC and non-invasive monitor

CONTACTS AND LOCATIONS:
Overall Officials: Katherine H Jelliffe, MD, Principal Investigator — UTMB; Antonio F Saad, MD, Study Director — UTMB
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No